CLINICAL TRIAL: NCT04038320
Title: Demonstration Project on Assessment of Simplified Antiviral Treatment Strategy for Hepatitis C in Ukraine
Brief Title: Simplified Antiviral Treatment Strategy for Hepatitis C in Ukraine
Status: Completed | Type: Observational
Sponsor: Right to Care (Other)
Collaborators: All Ukrainian Network of PLHA (Unknown); Public Health Center of MOH Ukraine (Unknown); Alliance for the Public's Health (Other); Boston University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: EQUIPHCV02-UKR
Record Dates: First submitted 2018-07-04; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; HIV; Key Population
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dry blood spots(DBS) collected at baseline, 4, 8, 12 and 24 weeks for viral load and resistance testing will be determined where indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCV infected patients: All HCV infected confirmed by HCV RNA,
  Interventions: Drug: Sofosbuvir/ledipasvir (SOF/LDV)

INTERVENTIONS:
Drug: Sofosbuvir/ledipasvir (SOF/LDV) — SOF/LDV (400mg/90mg) orally once daily with or without food in the morning and will receive treatment for a duration of 12 weeks.
  In addition, Ribavirin weight-based (1000 mg for patients <75 kg and 1200 mg for those ≥75 kg) administered orally in two divided doses with food for Genotype 3 patients.

SUMMARY:
The project will evaluate cost and treatment outcomes of a simplified Hepatitis C Virus (HCV) testing, treatment and care model integrated with HIV testing and treatment among key affected populations in Ukraine.

DETAILED DESCRIPTION:
Affected populations will be screened for HCV and HIV and those HCV positive treated with direct with direct acting anti-HCV agents (DAAs), a fixed-dose combination of sofosbuvir/ledipasvir (SOF/LDV) for 12 weeks with or without weight-based ribavirin. Before and after completion of the treatment course viral load assessments will be undertaken using low-cost laboratory monitoring for comparison to standard HCV viral load measurement. Up 800 patients enrolled on treatment will be followed up at 4, 8, 12 and 24 weeks when Sustained Viral Response (SVR) will be determined. Safety monitoring will be undertaken at applicable visits for those on Ribavirin and all adverse events will be reported based on Good Clinical Practice (GCP). In addition to assessing cost outcomes, the project will assess HCV treatment efficacy in terms of SVR at 12 weeks after end of treatment ( defined as undetected HCV RNA or less than lower limit of detection), compare the cost of low cost viral assay platforms to standard of care, assess rates of ART initiation and virologic suppression of HIV-infected persons within the simplified HCV treatment model and impact of HIV co-infection in participants on the HCV treatment outcome of SVR12. The project will be conducted at 2 treatment sites in Kiev.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness of participant to provide informed consent.
2. Attribution to one of the key population groups: People Who Inject Drugs (PWID), medication assisted treatment (MAT) participants, Commercial Sex Workers (CSW) or Men Having Sex with Men (MSM). Documentation of attribution to one of the key population groups will be done through applying Case Reporting Form "Risks Assessment" and "Substance Use and Alcohol Consumption". Additionally, medical record of substance use can be collected
3. Men and women age 18 years.
4. Active HCV infection as defined by detectable serum or plasma HCV RNA at any time prior to study entry. Documentation may be obtained from medical records if available. If no medical records on HCV infection are available, HCV infection must be confirmed by a detectable HCV RNA PCR prior to project entry.
5. Allowed HCV treatment history:

   1. HCV treatment naïve defined as not having been previously treated for Hepatitis C infection with any medications approved for the treatment of HCV in any country.
   2. HCV treatment experienced with interferon with or without ribavirin only (no prior DAA treatment, although they will be followed).
6. Hepatitis B status must be documented by hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), and hepatitis B core antibody (HBcAb) testing. Participants with positive hepatitis B surface antigen (HBsAg+) must be on an active HBV regimen at study entry.
7. HIV-1 infection status must be documented as either absent or present, as defined below:

   1. Absence of HIV-1 infection, as documented by rapid HIV test or HIV-1 enzyme immunoassay (ELISA) test kit, within 60 days prior to entry.

      OR
   2. Presence of HIV-1 infection, documented by rapid HIV test or HIV-1 ELISA test kit at any time prior to entry and confirmed by a second antibody test by a method other than the initial rapid HIV and/or ELISA, or by HIV-1 antigen or plasma HIV-1 RNA viral load.

      OR
   3. HIV-1 infection confirmed by medical documentation as participant is registered in care at AIDS Center and receiving or preparing to initiate ARV treatment.
8. Participants who are assigned to receive ribavirin as part of the treatment protocol must have haemoglobin ≥110 g/L
9. For females of reproductive potential, a negative urine pregnancy test (urine -HCG with a sensitivity of <25 mIU/mL) within 48 hours prior to project entry must be documented.
10. Male and female participants who are able to impregnate or become pregnant (ie, of reproductive potential) and are participating in sexual activity that could lead to pregnancy must agree to practice contraception/birth control as indicated below or agree to not participate in a conception process while on treatment with ribavirin through at least 12 weeks post-treatment.

Note: Acceptable contraception/birth control for this project includes one of the following methods:

* condoms (male or female) with a spermicide
* diaphragm or cervical cap with spermicide
* hormonally impregnated intrauterine device (IUD)
* non-hormonally impregnated IUD in conjunction with spermicide
* Hormone-based therapy

Exclusion Criteria

1. Child-Pugh Score corresponding to Class B or C (decompensated cirrhosis). This requires assessment for encephalopathy and ascites, as well as measurement of serum bilirubin, albumin, and international normalized ratio (Prothrombin time). For Child's cirrhosis severity calculator on the following link can be used: http://www.hepatitisc.uw.edu/page/clinical-calculators/ctp . Patients with decompensated cirrhosis and advanced liver disease will not be included to the treatment program, but they will remain under observation and will receive medical care within routine medical practice of the healthcare facility in such clinical cases.
2. Breastfeeding or pregnancy. Pregnant or breastfeeding woman will be documented and provided access to HCV treatment after resolution of pregnancy and breastfeeding.
3. Known allergy/sensitivity or any hypersensitivity to components of drug(s) or their formulation.
4. Active tuberculosis (TB) infection. Given the high TB prevalence in Ukraine, every candidate should be screened for TB signs/symptoms with further medical evaluation for active TB as indicated. In the case of proven active TB infection, the participant is ineligible for HCV treatment (due to the adverse drug interaction of SOF/LDV and rifampicin) but will be followed and offered enrolment when they complete treatment with rifampicin.
5. Renal impairment defined as estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 or end-stage renal disease receiving dialysis as treatment with SOF/LDV is contraindicated (https://www.mdcalc.com/mdrd-gfr-equation). The participant may be rescreened if the renal function improves. Patients with worse renal impairment will not be treated but will be followed and will recive medical aid within routine medical practice of the healthcare facility where project is implemented
6. Prior treatment with any HCV Direct Acting Agents (DAA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are HCV treatment naïve or experienced (pegylated interferon [PegIFN] and ribavirin [RBV] only), HCV-infected with genotype 1, 2, 3, 4, 5 or 6, men and women aged 18 years or older, with or without HIV-1 co-infection, representatives of key populations (PWID, CSW, MSM) and their partners. Participants with compensated cirrhosis or Hepatitis B will be eligible for HCV treatment. Patients with decompensated liver cirrhosis or prior treatment with HCV DAAs will not be eligible for treatment. HCV-infected patients who are not eligible for HCV treatment will be eligible for an observation arm.
Sampling Method: Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Estimated cost of HCV screening per patient screened and per case identified and the cost per successfully treated patient for HCV mono-infected and co-infected participants | Two years. This will be after data on Viral load response is complete.
  The average cost to the provider per patient achieving SVR-12 will be estimated, as will the average cost per other outcomes achieved, such as per patient screened and per patient remaining in care by other specified endpoints, stratified by HIV status and by any other important patient or site characteristics that are identified as drivers of cost. The investigators will also estimate the average cost to "produce" a successful outcome (SVR-12), which is the ratio of total costs for the intervention for the entire sample enrolled to the number of patients achieving the primary outcome. This latter estimate captures the costs incurred for patients who do not have successful outcomes and thus relates resource utilization to health outcomes.
Sustained Viral Response | 24 weeks ( 12 weeks post treatment)
  This will be the main treatment outcome of all patients initiated on treatment. Baseline viral load is done at entry with treatment initiated for those positive and eligible. Patients initiated on treatment will be assessed for viral load response at 24 weeks ( 12 weeks post treatment). This will also help in development of a Care cascade model for HCV testing, treatment and SVR12 in key populations co-infected with HIV/HCV, HIV/HCV/HBV, HBV/HCV and HCV mono-infected.

SECONDARY OUTCOMES:
HCV genotype | At baseline
  HCV genotype will be determined at entry for all patients.
HCV subtype | Baseline
  All genotypes will be subtyped once
Validity of Cepheid Gene-Xpert in monitoring SVR12 | Testing done and baseline and 24 weeks
  150 patients will be evaluated for HCV viral load at entry and exit comparing Cepheid Gen-Xpert and Real time PCR using Ampliscence platform.
HIV viral load among HCV/HIV co-infected patients | HIV Viral load at 24 weeks ( 12 weeks post HCV treatment)
  HCV/HIV co-infected patients will be on treatment at the time of HCV treatment initiation but those not on ART will be initiated and will assess rates of ART initiation and virologic suppression of the HIV infected within the simplified HCV testing and treatment model
Reliability of Cepheid Gene-Xpert in monitoring SVR12 | Testing done and baseline and 24 weeks
  Cepheid Gen-Xpert and Real time PCR using Ampliscence platform.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Sanne, MBBCH, FRCP, Study Chair — Right to Care; Svetlana Antonyak, MD, Principal Investigator — Hepatitis and HIV-infection of Institute of Epidemiology and Infectious Diseases of L.V. Gromashevskiy of NAMS of Ukraine; Tetiana Benard, MA, Principal Investigator — Right to Care, Ukraine; Charles Chasela, PhD, Study Director — Right to Care
Locations (2):
- Ukraine (2):
  - Clinic of the Institute of Epidemiology and Infectious Diseases, National Academy of Medical Sciences of Ukraine, Kiev
  - Kyiv City Clinical Hospital #5, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: One to two years after completion of the study
Access Criteria: Based on a concept submitted, reviewed and accepted

REFERENCES:
- [Result] Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol. 2014 Nov;61(1 Suppl):S45-57. doi: 10.1016/j.jhep.2014.07.027. Epub 2014 Jul 30. PMID 25086286
- [Result] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Result] Jaenisch T, Junghanss T, Wills B, Brady OJ, Eckerle I, Farlow A, Hay SI, McCall PJ, Messina JP, Ofula V, Sall AA, Sakuntabhai A, Velayudhan R, Wint GR, Zeller H, Margolis HS, Sankoh O; Dengue in Africa Study Group. Dengue expansion in Africa-not recognized or not happening? Emerg Infect Dis. 2014 Oct;20(10):e140487. doi: 10.3201/eid2010.140487. PMID 25271370
- [Result] Lazarus JV, Sperle I, Maticic M, Wiessing L. A systematic review of Hepatitis C virus treatment uptake among people who inject drugs in the European Region. BMC Infect Dis. 2014;14 Suppl 6(Suppl 6):S16. doi: 10.1186/1471-2334-14-S6-S16. Epub 2014 Sep 19. PMID 25252742
- [Result] Feld JJ, Jacobson IM, Hezode C, Asselah T, Ruane PJ, Gruener N, Abergel A, Mangia A, Lai CL, Chan HL, Mazzotta F, Moreno C, Yoshida E, Shafran SD, Towner WJ, Tran TT, McNally J, Osinusi A, Svarovskaia E, Zhu Y, Brainard DM, McHutchison JG, Agarwal K, Zeuzem S; ASTRAL-1 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. N Engl J Med. 2015 Dec 31;373(27):2599-607. doi: 10.1056/NEJMoa1512610. Epub 2015 Nov 16. PMID 26571066
- [Result] Gane EJ, Hyland RH, An D, Svarovskaia E, Pang PS, Brainard D, Stedman CA. Efficacy of ledipasvir and sofosbuvir, with or without ribavirin, for 12 weeks in patients with HCV genotype 3 or 6 infection. Gastroenterology. 2015 Nov;149(6):1454-1461.e1. doi: 10.1053/j.gastro.2015.07.063. Epub 2015 Aug 7. PMID 26261007
- See also: Over 5% of Ukrainians are infected with hepatitis C. 2016 — http://www.aph.org.ua/en/news/over-5-of-ukrainians-are-infected-with-hepatitis-c
- See also: EASL Recommendations on Treatment of Hepatitis C 2016. 2016 — http://www.easl.eu/research/our-contributions/clinical-practice-guidelines/detail/easl-recommendations-on-treatment-of-hepatitis-c-2016